CLINICAL TRIAL: NCT04491149
Title: The Ability of Virtual Reality in Anxiety and Pain Reduction in Women Undergoing Amniocentesis or Feticide
Brief Title: Study on the Ability of Virtual Reality Glasses in Anxiety and Pain Reduction in 50 Women Undergoing Amniocentesis or Feticide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #0182-19
Record Dates: First submitted 2020-06-14; First posted 2020-07-29 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-05

CONDITIONS: Anxiety Acute; Amniocentesis; Foeticide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women using virtual glass during amniocentesis/foeticide (Experimental)
  Interventions: Device: virtual reality glasses
- women undergoing amniocentesis/foeticide (No Intervention)

INTERVENTIONS:
Device: virtual reality glasses — In the intervention arm, women undergoing amniocentesis/foeticide will use virtual reality glasses during the procedure.
  Arms: women using virtual glass during amniocentesis/foeticide

SUMMARY:
Both amniocenteses and especially feticide are procedures that incorporate both anxiety and pain. As anxiety and pain can be reduced when using a distraction, The investigators speculate that the use of virtual reality glasses during these procedures will elevate both anxiety and pain.

The investigators will examine this hypothesis by comparing two groups of participants who undergo amniocentesis or feticide, one group will undergo the procedure while using virtual reality glasses and the other without the use of the glasses.

ELIGIBILITY:
Inclusion Criteria: Pregnant women undergoing amniocentesis/foeticide who will sign an informed consent form

-

Exclusion Criteria:

* Women younger than 18 years
* Twin pregnancies
* Women with vertigo

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | Up to one hour before the procedure
  Spielberger's State-Trait Anxiety Inventory
Anxiety level | Up to one hour after the procedure
  Spielberger's State-Trait Anxiety Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf ha Rofeh, MC, Zrifin, Israel